CLINICAL TRIAL: NCT02680782
Title: A Phase 1 Study Comparing Once-Daily vs. Twice-Daily Dosing of X4P-001 in Healthy Volunteers
Brief Title: A Study Comparing Once-Daily vs. Twice-Daily Dosing of X4P-001 in Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: X4 Pharmaceuticals (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: X4P-001-REGA
Record Dates: First submitted 2016-02-04; First posted 2016-02-12 (Estimated); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Healthy
Keywords: Healthy Volunteers; Comparison; Once-Daily; Twice-Daily; X4P-001
MeSH Terms: interventions — mavorixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- X4P-001 QD (Experimental): Subjects will receive study drug in two dosing periods. In this arm subjects will receive drug once daily in the first period, followed by twice daily in the second dosing period.
  Interventions: Drug: X4P-001
- X4P-001 BID (Experimental): Subjects will receive study drug in two dosing periods. In this arm subjects will receive drug twice daily in the first period, followed by once daily in the second dosing period.
  Interventions: Drug: X4P-001

INTERVENTIONS:
Drug: X4P-001 — 100 mg capsules, administered orally for 10 days either as 200 mg BID or 400 mg QD. Subjects will be randomized to determine if they will receive the drug QD or BID in the first dosing period.
  Other Names: AMD11070

SUMMARY:
This study will evaluate the safety, tolerability and pharmacokinetics of X4P-001 administered as 200 mg twice daily compared with 400 mg once daily.

This study will also assess the pharmacodynamic effects of X4P-001 administered as 200 mg twice daily compared with 400 mg once daily on levels of circulating white blood cells (total and by cell type).

DETAILED DESCRIPTION:
This study will be conducted in 15 healthy volunteers at a clinical research unit located in Daytona Beach, Florida. Screening will be done within 35 days prior to the first dose of study drug (first Dosing Period). Each subject will complete two 10-day Dosing Periods, one using once daily dosing and the other twice daily dosing. The interval between the Dosing Periods will be 7 to 17 days. Patients will be randomly assigned to which regimen is administered the first Dosing Period. Safety laboratory tests will be performed at screening, and prior to and after each Dosing Period. End-of-Study (EOS) visit, the final study event, will be performed 14 to 21 days after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 and 65 years of age, inclusive.
2. Have signed the current approved informed consent form.
3. For women of childbearing potential, (a) agree to use effective contraceptive methods from screening, through the study, and for at least 4 weeks after the last dose of study drug; and (b) have a negative pregnancy test (serum or urine) at screening and on Day -1 prior to each Dosing period.
4. For men, agree both to (a) use effective contraceptive methods and (b) abstain from donating sperm, from admission to the in-residence unit prior to the first Dosing Period, through the study, and for at least 4 weeks after the last dose of study drug.
5. Be willing and able to comply with this protocol.

Exclusion Criteria:

1. Is an employee of the Phase 1 unit or an immediate family member of an employee.
2. Has a BMI <18.0 or >30.0.
3. Has a history of hypersensitivity or allergy to any drug compound, food or other substance assessed as significant by the Investigator.
4. Has a history or presence of any medical condition capable of altering absorption, metabolism or elimination of drugs (history of routine cholecystectomy is permitted).
5. Has alcohol intake exceeding 21 units per week for males or 14 units per week for females, where 1 unit = 12 oz (360 mL) beer, 5 oz (150 mL) wine, or 1.5 oz (45 mL) distilled spirits.
6. Has within the past 12 months used illicit drugs.
7. Has within the past 6 months been a smoker or used tobacco or nicotine replacement products.
8. Is within 6 months post-partum or termination of a pregnancy.
9. Has within the past 30 days or 5 half-lives, whichever is longer, participated in any other clinical trial involving an investigational treatment.
10. Has within the past 30 days had an acute medical illness, including an active infection.
11. Has within the past 30 days donated more than 500 mL of blood.
12. Has within the past 30 days, or is scheduled to have while participating in the study, surgery requiring general anesthesia.
13. Has within the past 30 days, or is scheduled to have while participating in the study, any immunizations.
14. Has within the past 14 days been nursing.
15. Has within the past 14 days donated plasma.
16. Has within the past 14 days used any prescription or over the counter medications, unless deemed acceptable by the Investigator.
17. Has positive urine or serum test for drugs of abuse or for cotinine.
18. Has positive serologic laboratory tests:

    * Human immunodeficiency virus (HIV-1 or -2)
    * Hepatitis C virus (HCV)
    * Hepatitis B virus (HBV)
19. Has confirmed abnormal safety laboratory tests representing CTCAE Grade 2 or higher. Subjects with Grade 1 abnormalities may be enrolled with the approval of the Investigator and the Sponsor.
20. Has insufficient venous access to permit the scheduled blood sampling.
21. Has any other medical or personal condition or finding that, in the opinion of the Investigator, may potentially compromise the safety or compliance of the subject, or may preclude the subject's successful completion of the clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-01-12 (Actual); Primary Completion 2016-02-28 (Actual); Study Completion 2016-02-28 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events (safety and tolerability) in subjects administered X4P-001 200 mg twice daily compared with 400 mg once daily. | Up to 14 to 21 days post-last dose
  Safety assessments include ongoing monitoring of adverse events, ongoing monitoring of concomitant medications and regulatory scheduled vital signs, physical examinations and laboratory tests (hematology, clinical chemistry, urinalysis and coagulation).
Maximum Plasma Concentration (Cmax) of X4P-001 administered as 200 mg twice daily compared with 400 mg once daily. | Up to 48 hours post-dose
  Cmax data will be collected to determine the pharmacokinetics of X4P-001 administered as 200 mg twice daily and 400 mg once daily.
Area under the curve (AUC) of X4P-001 administered as 200 mg twice daily compared with 400 mg once daily. | Up to 48 hours post-dose
  AUC data will be collected to determine the pharmacokinetics of X4P-001 administered as 200 mg twice daily and 400 mg once daily.
Minimum Plasma Concentration (Cmin) of X4P-001 administered as 200 mg twice daily compared with 400 mg once daily. | Up to 48 hours post-dose
  Amin data will be collected to determine the pharmacokinetics of X4P-001 administered as 200 mg twice daily and 400 mg once daily.

SECONDARY OUTCOMES:
To assess the pharmacodynamic effects of X4P-001 administered as 200 mg twice daily compared with 400 mg once daily on levels of circulating white blood cells (total and by cell type). | Up to 48 hours post-dose
  Whole blood samples will be obtained for PD studies concurrently with the PK samples. PD will be assessed via complete blood counts (CBC) with differential.
To assess the pharmacodynamic effects of X4P-001 administered as 200 mg twice daily compared with 400 mg once daily on levels of circulating mononuclear cell phenotypes by cell surface markers. | Up to 48 hours post-dose
  Whole blood samples will be obtained for PD studies concurrently with the PK samples. PD will be assessed via complete blood counts (CBC) with differential.

CONTACTS AND LOCATIONS:
Overall Officials: Lu Gan, MD, PhD, Study Director — X4 Pharmaceuticals, Inc.
Locations (1):
- Covance CRU, Inc., Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No